CLINICAL TRIAL: NCT05972317
Title: Generating a Stool Microbiome-based Diagnostic for IBS (Irritable Bowel Syndrome) Patients in Low-FODMAP Treated and Untreated IBS Patients
Brief Title: The Stool Microbiome of Treated and Untreated IBS (Irritable Bowel Syndrome) Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1914-4
Record Dates: First submitted 2023-03-02; First posted 2023-08-02 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-02

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-IBS (No Intervention): Participants which are not suffering from IBS symptoms.
- IBS -low FODMAP (Experimental): individuals that are diagnosed with IBS according to Rome IV criteria
  Interventions: Other: Low FODMAP dietary regimen
- FODMAP graduates (No Intervention): Individuals who have practiced a low-FODMAP diet in the past

INTERVENTIONS:
Other: Low FODMAP dietary regimen — intervention will include a guidance by a clinical dietitian about low FODMAP diet
  The FODMAP diet has three phases:
  1. Elimination - Avoidance from high-FODMAP foods (2-6 weeks)
  2. Reintroduction -Structured challenges of specific food groups each time (6-8 weeks).
  3. Maintenance - personalized diet, according to the response in step 2.
  Arms: IBS -low FODMAP

SUMMARY:
Irritable bowel syndrome (IBS) is considered the most common gastrointestinal disorder in humans, with an estimated global prevalence of 11%-20% of all humans. Alterations in the gut microbiome are at the center of IBS, and microbiome-induced volatile metabolites in response to dietary exposures is believed to drive a downstream impact on susceptible hosts, thereby driving the disease. However, the characteristics and functions of these metabolites remain unknown to date. The two main mechanisms invoking IBS development and flares include 1) an increase in luminal water content due to malabsorption of small molecules and 2) incrementation of colon gas production generated by the fermentation of small molecules by gut bacteria.Yet to date, a person-specific elucidation of the specific small molecules and bacteria driving IBS, and their downstream effects on the human gut epithelium remain unknown.

Over the past years, it became evident that dietary regimes, and their interactions with the intestinal microbiome, are at the center of IBS symptom generation and alleviation. The most widely used dietary intervention is a highly restrictive diet, the low-Fermentable Oligo-saccharides Di-saccharides Mono-saccharides And Polyols (FODMAP) diet, based on avoidance of multiple food items that contain available fermentable molecules.

The low-FODMAP diet remains an effective line of treatment for IBS patients, yet due to its complexity and unhealthy nature, it remains a last line of treatment and fails to impact the majority of IBS patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Age - 18-70

Exclusion Criteria:

* Consumption of antibiotics 2 months prior to the first day of the experiment.
* Consumption of probiotic supplements 1 month prior to the first day of the experiment.
* Type 1 or type 2 diabetes diagnosis.
* Pregnancy, fertility treatments, breastfeeding 3 months prior to the first day of the study.
* Chronic disease - to the discretion of the study doctor.
* Cancer and recent anticancer treatment.
* Psychiatric disorders - to the discretion of the study doctor.
* IBD (inflammatory bowel diseases).
* Alcohol or substance abuse.
* BMI > 35.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
IBS-SSS - irritable bowel syndrome severity score system questionnaire | 1 week
  Severity of symptoms as they are scored in the Rome IV IBS-SSS 75 to <175 to indicate mild IBS, 175 to <300 as moderate, and >300 as severe
IBS-QOL questionnaire - irritable bowel syndrome quality of life questionnaire | 1 week
  Quality of life scores from the Rome IV IBS-QOL 0-100 scale for ease of interpretation with higher scores indicating better IBS specific quality of life

SECONDARY OUTCOMES:
Stool microbiome differences between the study arms - using fecal samples of participants | 3 months
  Analysis of stool samples of the different study arms - using shot-gun metagenomics to asses type of microbiota pre and post low-FODMAP diet.

CONTACTS AND LOCATIONS:
Overall Officials: Eran Elinav, Prof, Principal Investigator — Weizmann Institute of Science
Locations (1):
- Weizmann institute of science, Rehovot, Israel, Israel